CLINICAL TRIAL: NCT03115593
Title: Compare the Performance of Targeted Biopsy Versus Aspiration Biopsy With a Pipette for the Diagnosis of Endometrial Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of human ressources
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Andre Nazac, Head of clinic, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-Hystocor
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Endometrial Cancer
Keywords: hysteroscopy; pipette; biopsy; endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- postmenopausal patients with metrorrhagia (Experimental): Postmenopausal patients with metrorrhagia and endometrial hypertrophy defined by an endometrium ticker than 3 mm (ultrasound result).
  The threshold choice of 3 mm was chosen according to a recent review of the literature to limit the risk of false negatives for cancer.
  Interventions: Procedure: Blind biopsy with a pipette; Procedure: Targeted biopsy using hysteroscopy

INTERVENTIONS:
Procedure: Blind biopsy with a pipette — Patients willing to participate to the study will benefit from a double biopsy. The first biopsy will be a blind biopsy performed by aspiration with a Cornier pipette.
Procedure: Targeted biopsy using hysteroscopy — During the same consultation, patients will benefit from a diagnostic hysteroscopy with vaginoscopy and saline (allowing a wash of the debris caused by the pipette biopsy), using a rigid hysteroscope of 4.3 mm equipped with an operator channel allowing the passage of a biopsy tong.

SUMMARY:
Endometrial cancer is the most common pelvic gynecological cancer in so-called developed countries, with 320,000 new cases annually, including more than 1,500 in Belgium. It preferentially affects postmenopausal women. Overall survival at 5 years is 76% but is 95% for early forms, which represent more than 70% of diagnoses. The main risk factors are obesity, diabetes and tamoxifen intake for breast cancer, which explains the increasing incidence. Half a million new annual cases are expected in 2035.

The main symptom is postmenopausal metrorrhagia.Among these women, the prevalence of the disease is estimated between 10 and 15%. Currently the recommendations are to make an evaluation by endovaginal ultrasound followed by an endometrial biopsy. The histological type is the main predictor of the severity of the disease and acts as guideline for the treatment.It is therefore essential to have precise biopsy results before starting therapeutic management.

The most widely used technique is the blind biopsy by aspiration using a pipette because it is inexpensive, easy, without any specific equipment. However, recent studies showed that this technique has a poor sensitivity in the target population of postmenopausal women. Other studies have shown that targeted biopsies under hysteroscopic control could have a much higher sensitivity.

The main objective of this study is thus to compare the performance of the targeted biopsy under hysteroscopy to the performance of the biopsy by aspiration with a pipette, for the diagnosis of endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal patient.
* patient with postmenopausal metrorrhagia and endometrial hypertrophy defined by an endometrium ticker than 3 mm (ultrasound result)

Exclusion Criteria:

* patients undergoing hormone replacement therapy for menopause (THM). This treatment may be the cause of benign bleeding in post menopause.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Histological result | 6 months
  Histological result (histological type and grading if cancer is diagnosed, according to the FIGO 2009 classification).

CONTACTS AND LOCATIONS:
Overall Officials: André Nazac, MD, Principal Investigator — CHU Brugmann
Locations (4):
- Belgium (3):
  - CHU Brugmann, Brussels
  - Hôpitaux Iris Sud - Site Ixelles, Brussels
  - CHR Citadelle, Liège
- Hôpital Bicêtre, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No